CLINICAL TRIAL: NCT02702856
Title: Clinical Validation of a Urinary Exosome Gene Signature in Men Presenting for Suspicion of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Exosome Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECT2014-001A
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Gleason Grade; Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Prospectively collect approximately 25-40mL of random, non-DRE, non catheter urine, in a standard, reduced size, clinical capture vessel.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Men screened for prostate cancer
  Interventions: Other: ExoIntelliScore Prostate

INTERVENTIONS:
Other: ExoIntelliScore Prostate

SUMMARY:
Validate a non-DRE exosome gene expression test, with an NPV >/= 90% certainty, will exclude the presence of high gleason grade/ score (>/=7) prostate cancer in a prostate needle biopsy.

DETAILED DESCRIPTION:
The purpose of this multi-center clinical study is to determine the association of an Exosome Urine Test score with the presence of high Gleason grade / score (GS>/=7) prostate cancer on a prostate needle biopsy and validate the assay's performance characteristics in men presenting to their urologist with or without a previous negative biopsy, and recommended for an initial or subsequent biopsy. The results of this study are to support the use of this assay as a laboratory developed test. A secondary objective is to develop an assay that accurately predicts the presence of any Gleason grade prostate cancer in men at risk for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male, >50 years of age with a clinical suspicion for prostate cancer based in part on an elevated PSA (limit range: 2.0 - 20 ng/ mL), and or suspicious DRE, with or without the clinical history of a single prior negative biopsy, and who have been recommended for a repeat and or first time biopsy.
2. The subject must be able to comprehend and sign an approved informed consent form and other applicable study documents.

Exclusion Criteria:

1. Use of medications or hormones that are known to affect serum PSA levels within 3-6 months of study enrollment.
2. Clinical symptoms of urinary tract infection (including prostatitis) at the time of enrollment.
3. History of prostate cancer.
4. History of invasive treatments for benign prostatic hypertrophy (BPH) or lower urinary track symptoms within 6 months of study enrollment.
5. Medical history or concurrent illness that the investigator considers sufficiently serious to interfere with the conduct, completion or results of this trial, or constitutes an unacceptable risk to the subject.
6. Participation in pharmaceutical or treatment related clinical study within 6 months of study enrollment. Exception: Trials for non-prostate conditions may be acceptable, with approval by the investigator and Sponsor.
7. No known hepatitis (all types) and/or HIV documented in patient's medical record.
8. Patients with history of concurrent renal/bladder tumors within 6 months of study enrollment.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Correlate an exosome gene expression signature with the presence or absence of high grade prostate cancer in the prostate needle biopsy. | one year
  Validate various thresholds utilizing the exosome RNA gene signature to stratify patients based on the likelihood of having any Gleason pattern 4 disease present within the biopsy (or when available the prostatectomy specimen surgical pathology report) for first time biopsy patients in the PSA gray zone of 2.0-10 ng/mL. In our earlier cohort analyses and in the literature there is an expected 20-25% of patients who will present with Gleason score >/=7 and the prevalence of a dominant Gleason 4 varies considerably dependent upon studies from 17-30%.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Tun, Study Director — Exosome Diagnostics, Inc.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kretschmer A, Tutrone R, Alter J, Berg E, Fischer C, Kumar S, Torkler P, Tadigotla V, Donovan M, Sant G, Skog J, Noerholm M. Pre-diagnosis urine exosomal RNA (ExoDx EPI score) is associated with post-prostatectomy pathology outcome. World J Urol. 2022 Apr;40(4):983-989. doi: 10.1007/s00345-022-03937-0. Epub 2022 Jan 27. PMID 35084544